CLINICAL TRIAL: NCT01671410
Title: A Randomized, Open Label Clinical Trial of Buprenorphine in the Treatment of Neonatal Abstinence Syndrome in Infants With In Utero Exposure to Benzodiazepines or Are Breastfeeding
Brief Title: Buprenorphine for Treatment of Neonatal Abstinence Syndrome in Infants With In Utero Exposure to Benzodiazepines
Acronym: MOPPlus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12D.398
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: Neonatal Abstinence Syndrome; buprenorphine; morphine; benzodiazepine
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Morphine; Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sublingual buprenorphine (Experimental): Initial daily dose: 15.9 mcg/kg/day; Initial unit dose: 5.3 mcg/kg q8 hours; Maximum daily dose: 60 mcg/kg/day; Up-titration rate: 25%; Weaning rate: 10%; Cessation Dose: Within 10 or 20% of starting dose
  Interventions: Drug: sublingual buprenorphine
- oral morphine (Active Comparator): Initial daily dose: 0.4 mg/kg/day; Initial unit dose: 0.07 mg/kg q 4 hours; Maximum daily dose: 1.25 mg/kg/day; Up-titration rate: 20%; Weaning rate: 10%; Cessation Dose: 0.025 mg/kg q 4 hours
  Interventions: Drug: oral morphine

INTERVENTIONS:
Drug: oral morphine — Oral morphine for the treatment of neonatal abstinence syndrome
  Other Names: morphine
  Arms: oral morphine
Drug: sublingual buprenorphine — Sublingual buprenorphine for the treatment of neonatal abstinence syndrome
  Other Names: buprenex
  Arms: sublingual buprenorphine

SUMMARY:
The opioid neonatal abstinence syndrome (NAS) is a condition of withdrawal symptoms after utero exposure to opioids. Sublingual buprenorphine shows promise as a new treatment in NAS. This trial will investigate the safety and tolerability of sublingual buprenorphine in infants exposed to both opioids and benzodiazepines in utero or with exposure of opioids in those who are breastfeeding.

DETAILED DESCRIPTION:
Infants with in utero exposure to opioids often require therapy with morphine for an extended period. In a clinical trial, sublingual buprenorphine reduced this treatment period by ~30%. However, infants with both opioid and benzodiazepine exposure were not included in the trial. This study will test the safety and tolerability of sublingual buprenorphine in infants with in utero exposure to benzodiazepines or who are breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 37 weeks gestation
2. Exposure to opioids in utero
3. Demonstration of signs and symptoms of neonatal abstinence syndrome requiring treatment
4. Exposure to benzodiazepines in utero and/or receiving breast milk. Benzodiazepine use is defined as maternal use in the past 30 days, and/or receipt of benzodiazepines by prescription (as determined by self-report or intake urine) by the mother 30 days prior to birth.

Exclusion Criteria:

1. Major congenital malformations and/or intrauterine growth retardation defined as birth weight <2200 gm
2. Medical illness requiring intensification of medical therapy. This includes, but is not limited to suspected sepsis requiring antibiotic therapy.
3. Hypoglycemia requiring treatment with intravenous dextrose
4. Bilirubin >20 mg/dL (The need for phototherapy is not exclusionary)
5. Seizure activity or other neurologic abnormality

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Length of treatment | Patients will be followed for the duration of hospital stay, an expected average of 5 weeks
  This endpoint will compare length of treatment (in days) using sublingual buprenorphine or oral morphine solution.

SECONDARY OUTCOMES:
Length of hospitalization | Patients will be followed for the duration of hospital stay, an expected average of 5 weeks
  This endpoint will compare length of stay (in days) using sublingual buprenorphine or oral morphine
Number of patients requiring supplemental phenobarbital treatment | Patients will be followed for the duration of hospital stay, an expected average of 5 weeks
  This endpoint will compare requirement number of patients who require use of supplemental phenobarbital for treatment of NAS
Number of participants with adverse events as a measure of safety and tolerability | Patients will be followed for the duration of hospital stay, an expected average of 5 weeks
  Adverse events will be collected, graded by severity, and assessed for causality referent to study drug.

OTHER OUTCOMES:
Feeding patterns | Patients will be followed for the duration of hospital stay, an expected average of 5 weeks
  To compare the feeding patterns, weight gain, and incidence of feeding dysfunction in infants treated with sublingual buprenorphine and oral morphine for NAS
Respiratory Patterns | Patients will be followed for the duration of hospital stay, an expected average of 5 weeks
  To compare the respiratory patterns of infants receiving sublingual buprenorphine or morphine solution for the pharmacologic treatment of NAS after in utero exposure to opioids and benzodiazepines and/or postnatal breast milk.

CONTACTS AND LOCATIONS:
Overall Officials: Walter K Kraft, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States